CLINICAL TRIAL: NCT01898650
Title: MRI for Non-invasive Evaluation of Brain Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201208086
Record Dates: First submitted 2012-12-06; First posted 2013-07-12 (Estimated); Results first posted 2023-02-01 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Craniosynostosis
Keywords: craniosynostosis; sagittal synostosis; metopic synostosis; coronal synostosis; lambdoid synostosis
MeSH Terms: conditions — Craniosynostoses

STUDY DESIGN:
Intervention Model Description: individual participants will serve as their own controls by using affected and unaffected regions of the brain for paired analysis
Oversight: Data Monitoring Committee: No

ARMS (1):
- craniofacial abnormalities (Experimental): Subjects with craniosynostosis or other craniofacial abnormalities associated with ICP who will undergo an MR scan.
  Interventions: Other: MR scan

INTERVENTIONS:
Other: MR scan

SUMMARY:
Craniosynostosis is a birth defect that causes the bones on a baby's head to fuse together earlier than normal. This causes the baby to have an abnormally shaped head. These children are operated on to prevent or treat increased pressure on the brain, allowing for normal development. There is not good evidence of which children with craniosynostosis have increased pressure on the brain. Up to twenty patients with craniofacial abnormalities will be enrolled in this pilot study. The investigators will use a magnetic resonance scanner to obtain several measures of brain metabolism. The investigators will also obtain data which are markers of developmental delay.

The results will also be compared to age and gender matched data from children without craniofacial abnormalities.

There study hypothesis is that patients with craniofacial abnormalities associated with intracranial pressure will have decreased metabolic activity compared to control patients.

DETAILED DESCRIPTION:
The incidence of craniosynostosis is reported to be 1/2,000 births. Craniosynostosis is a birth defect that causes one or more sutures on a baby's head to close earlier than normal. The skull of an infant or young child is made up of bony plates that allow for growth of the skull. The borders at which these plates intersect are called sutures or suture lines. Early closing of a suture causes the baby to have an abnormally shaped head.

Original contributions by Dr. Paul Tessier along with technological advances (improved pediatric anesthesia, rigid fixation, resorbable plates, endoscopic techniques and distraction) have significantly advanced surgical treatment for these patients over the past 40 years.

Primary indication for operative treatment for patients with craniosynostosis is to prevent or treat increased intracranial pressure (ICP) and avoid neurological impairment. Increased ICP is thought to result from restricted space for brain growth caused by decreased cranial vault volume. A secondary surgical indication is normalization of head shape for cosmetic purposes.

Literature is limited on the relationship between craniosynostosis and ICP. The most widely reported study is by Renier and colleagues. In 75 patients preoperative ICP monitoring was performed using an epidural sensor. They identified ICP to be normal in one-third of the cases, obviously elevated in one-third, and borderline in one-third. When counseling patients, practitioners report a 13% rate of increased ICP for single suture synostosis and 42% for multiple suture synostosis. However, the authors used adult normative values for ICP (normal less than 10mmHg and elevated greater than 15mmHg). Normal ICP in children and infants has been identified to be closer to 6 mmHg.

Due to the invasiveness of the test, preoperative ICP monitoring is not routinely performed to decide if operative repair is required. Other indirect signs of increased intracranial pressure have been described (e.g., copper beaten appearance of the skull on plain film, papilledema, comparing intracranial volume to normative data), but are not reliable. Currently, the standard of care is to surgically treat all patients with craniosynostosis.

While it is not currently feasible to measure ICP directly, we may be able to indirectly study the effects of growth restriction on brain development. Metabolic consequences of direct mechanical stress and global cerebral ischemia in craniosynostosis have not been described. We aim to evaluate the prevalence of metabolic defects in craniosynostosis patients through the use of magnetic resonance (MR) imaging techniques.

Up to twenty patients with craniosynostosis or other abnormalities such as hydrocephaly which are associated with increased cranial pressure will be enrolled in this pilot study. The investigators will obtain several measures of cerebral metabolism preoperatively. MR spectroscopy (MRS) will be used to obtain concentrations of N-acetyl aspartate (NAA) and lactate. NAA is a highly sensitive marker of brain injury and the presence of lactate can indicate compromised metabolism. We will measure whole-brain oxygen extraction (OEF) using a magnetic field mapping approach. Elevated OEF is a key indicator of compromised perfusion. Cerebral blood flow (CBF) will be measured using an arterial spin labeling (ASL) sequence, which will allow direct measurement of perfusion deficiencies. We will also obtain functional connectivity data using an rfcMRI sequence, which is sensitive to developmental delay. Finally, a scanner sequence which measures CSF flow as a marker of intracranial pressure will also be performed.

The results will also be compared to deidentified age and gender matched normative data. These controls will be recruited in the plastic surgery clinic and/or deidentified data from normal subjects from another study will be used. The analysis for OEF and ASL data will be performed by Dr. Dustin Ragan and Dr. McKinstry at Washington University in St. Louis.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to the Plastic Surgery or Neurosurgery clinics with scheduled sedated MRI and abnormalities such as hydrocephalus (and possibly some patients to be used as controls who present to the clinic with no known skull or brain abnormalities)

Exclusion Criteria:

* history of abnormalities known to affect brain topology or function
* implants (e.g. pacemakers) that might rule out use of MR scanning.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2013-01-30 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamlesh Patel, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the beginning of 2013 (anticipated date) until September 2014 (anticipated date).
Groups:
- Craniofacial Abnormalities: Subjects with craniosynostosis or other craniofacial abnormalities associated with ICP who will undergo an MR scan.
  MR scan
Period: Overall Study
Arm/Group | Craniofacial Abnormalities
Started | 12 (12 were enrolled, beginning on 1/30/2013)
Scanned | 11
Completed | 11 (last subject scanned)
Not Completed | 1
Not completed — the subject would not lie still for imaging | 1

BASELINE CHARACTERISTICS:
Arm/Group | Craniofacial Abnormalities
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Blood Flow and Perfusion
Description: To be measured with both oxygen extraction fraction and arterial spin labeling to measure blood flow.
Time Frame: during the single MRI scan, approximately 30 - 45 minutes
Measure: Mean (Standard Deviation); unit: ml/min/100g
Arm/Group | Craniofacial Abnormalities
Number analyzed (Participants) | 6
ml/min/100g | 26.8 (5.6)
Statistical Analysis 1: Comparison: Craniofacial Abnormalities; Null hypothesis was that blood flow would be equivalent on the unaffected and affected sides; Test type: Superiority; p = 0.004, t-test, 1 sided — no adjustments for multiple comparisons were made. the threshold for significance was set a priori at 0.05

ADVERSE EVENTS:
Time Frame: during the single study visit, a 30 - 45 minute MRI scan
Arm/Group | Craniofacial Abnormalities
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

LIMITATIONS AND CAVEATS:
A primary limitation of this study is the small sample size and the variability between subjects with respect to their diagnosis and condition.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT01898650/Prot_SAP_000.pdf